CLINICAL TRIAL: NCT03603860
Title: Comparison of Continuous Blood Pressure Measurement Using the Non-invasive, Wireless Biobeat Monitor With an Invasive Arterial Line
Brief Title: Comparison of the Non-invasive Biobeat Device With an Invasive Arterial Line
Status: Completed | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Collaborators: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Other Study IDs: Biobeat001
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-01

CONDITIONS: Blood Pressure; Heart Diseases
Keywords: vital signs; blood pressure; cardiac surgery; non-invasive monitoring
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non-invasive monitoring — Comparing blood pressure measurement using the Biobeat non-invasive monitor to arterial line

SUMMARY:
In this clinical study the investigators will compare blood pressure measurements obtained using the non-invasive, continuous and wireless Biobeat monitoring device (a wrist watch or a patch configuration) to an invasive arterial line (radial or femoral) in 30 patients immediately after cardiac surgery, at the intensive care unit.

DETAILED DESCRIPTION:
The Biobeat non-invasive, continuous and wireless monitoring device is based on photoplethysmograph technology. It measures several vital signs, including blood pressure, stroke volume, pulse rate, pulse pressure, heart rate variability, respiratory rate, saturation, cardiac output, cardiac index, and more. The data is transmitted to Biobeat's application (in both Apple and Google Play), and is available on the individual's cellular phone, tablet, or as a full monitoring system in a hospital department. The aim of this study is to compare the Biobeat monitor with the invasive method of blood pressure measurement, an arterial line. The study population includes 30 patients undergoing cardiac surgery. As per local protocol, each one of the participants will come out from the operating room with an arterial line. Once in the intensive care unit, the investigators will attach the Biobeat non-invasive monitor (either wrist watch or a patch, these two configurations are identical in terms of the monitoring system), and monitor the participants for 4 hours. Though both methods are continuous, the investigators will record the vital signs every 15 minutes during the 4 hours of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients arriving immediately after cardiac surgery to the intensive care unit with an arterial line.

Exclusion Criteria:

* Refusal to participate
* Patients with no arterial line
* Pregnant women
* Individuals under the age of 18 years
* Patients with lack of judgment/mental illness
* Patients working in the Baruch Padeh Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients immediately after cardiac surgery arriving to the intensive care unit, and connected to an arterial line transducer. Usually the arterial line is left for 24 hours. Right after arrival and once connected to an arterial line, the participants will be connected to the Biobeat monitor (either wrist watch or a patch). Vital signs will be monitored for 4 hours, and recorded every 15 minutes, for comparison. After 4 hours, the Biobeat monitor will be disconnected.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Level of accordance between the Biobeat monitor and the arterial line | 4 hours per individual
  Comparing blood pressure measurements of the Biobeat device with those of the arterial line. Both systolic blood pressure and diastolic blood pressure will be assessed during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Kachel, MD, Principal Investigator — The Baruch Padeh Medical Center, Poriya, Israel
Locations (1):
- The Baruch Padeh Medical Center, Poriya, Tiberias, Lower Galilee, Israel

IPD SHARING:
Plan to Share IPD: Undecided
The investigators would probably share the results showing the level of agreement between the two measurement methods, but it will not be an individual data, rather the whole group, without any personal data included.

REFERENCES:
- [Derived] Eisenkraft A, Goldstein N, Ben Ishay A, Fons M, Tabi M, Sherman AD, Merin R, Nachman D. Clinical validation of a wearable respiratory rate device: A brief report. Chron Respir Dis. 2023 Jan-Dec;20:14799731231198865. doi: 10.1177/14799731231198865. PMID 37612250
- [Derived] Kachel E, Constantini K, Nachman D, Carasso S, Littman R, Eisenkraft A, Gepner Y. A Pilot Study of Blood Pressure Monitoring After Cardiac Surgery Using a Wearable, Non-invasive Sensor. Front Med (Lausanne). 2021 Aug 5;8:693926. doi: 10.3389/fmed.2021.693926. eCollection 2021. PMID 34422859